CLINICAL TRIAL: NCT06141252
Title: Benefit of Hypothermia in Out-of-hospital Cardiac Arrest Complicating Acute Myocardial Infarction
Brief Title: Benefit of Hypothermia in OHCA Complicating AMI
Acronym: Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, SungA Bae, Clinical Professor, Yonsei University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Door-to-cooling timing in OHCA
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Myocardial Infarction, Acute; Hypothermia Neonatal
Keywords: Out-Of-Hospital Cardiac Arrest; Acute myocardial infarction; Hypothermia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Myocardial Infarction; Hypothermia

STUDY DESIGN:
Intervention Model Description: The investigators aim to compare and evaluate the effects of therapeutic hypothermia versus standard care on clinical outcomes, such as survival rates and neurological function, in patients with out-of-hospital cardiac arrest complicating acute myocardial infarction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypothermia (Experimental): Patients admitted with out-of-hospital cardiac arrest and treated with hypothermia
  Interventions: Device: Hypothermia
- No hypothermia (No Intervention): Patients admitted with out-of-hospital cardiac arrest and treated without hypothermia

INTERVENTIONS:
Device: Hypothermia — Patients admitted with out-of-hospital cardiac arrest and treated with hypothermia
  Arms: Hypothermia

SUMMARY:
To determine the clinical effectiveness of hypothermia treatment in patients with out-of-hospital cardiac arrest complicating acute myocardial infarction.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a leading cause of mortality worldwide. Due to significant improvement in the management of patients with OHCA, an increasing number of initially resuscitated patients are being admitted to hospitals. Nevertheless, OHCA remains associated with a poor prognosis, with a survival rate of approximately 8.8% to hospital discharge. Moreover, international registry data have indicated that favorable neurological outcome at hospital discharge or 30 days after OHCA is only 2.8-18.2% across all registries.

The majority of adult cardiac arrest cases are associated with obstructive coronary artery disease. Thus, current guideline recommended that immediate angiography and primary revascularization in all patients with resuscitated cardiac arrest and ST-segment elevation on electrocardiography, and also in patients with resuscitated cardiac arrest without ST-segment elevation, but with high probability of acute coronary occlusion. However, even after prompt restoration of blood flow, a substantial proportion of patients with myocardial infarction (MI) experience extensive necrosis. The application of hypothermia in patients with acute MI focuses on the reducing energy consumption at cardiac level, a factor consistently linked to diminished infarction size in animal study. However, in a recent meta-analysis of randomized trials comparing different strategies for therapeutic hypothermia adjunctive to percutaneous coronary intervention (PCI) versus standard of care in patients with acute MI, faille to demonstrate clear benefit. It is important to note, however, these randomized trials were underpowered and as a results, they were unable to draw firm conclusions regarding the impact of therapeutic hypothermia.

Therefore, this study aimed to investigate the impact of therapeutic hypothermia on clinical outcomes in patients who underwent primary PCI for acute MI after OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest event

Exclusion Criteria:

* Arrest of non-cardiac origin
* Age < 18 years
* Did not received primary PCI
* Hypothermia before CAG
* Obey mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2925 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Death from any cause at hospital discharge | up to 30 days
  Death from any cause at hospital discharge

SECONDARY OUTCOMES:
Poor neurological outcomesat hospital discharge | up to 30 days
  Poor neurological outcomes, which was defined as a Glasgow-Pittsburge Cerebral Performance Category (CPC) value at hospital discharge. The investigators determined the neurological outcome according to Pittsburgh CPC, which is a scale on 1 to 5. 1 is e.g. good cerebral performance: conscious, alert, able to work, might have mild neurological or physiological deficit contrast to 5 which is brain death.

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Yongin Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yongin Severance Hospitall, Yonsei University College of Medicine, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker L, Gold LS, Eisenberg M, White L, Hearne T, Rea T. Ventricular fibrillation in King County, Washington: a 30-year perspective. Resuscitation. 2008 Oct;79(1):22-7. doi: 10.1016/j.resuscitation.2008.06.019. Epub 2008 Aug 6. PMID 18687513
- [Background] Berdowski J, Berg RA, Tijssen JG, Koster RW. Global incidences of out-of-hospital cardiac arrest and survival rates: Systematic review of 67 prospective studies. Resuscitation. 2010 Nov;81(11):1479-87. doi: 10.1016/j.resuscitation.2010.08.006. Epub 2010 Sep 9. PMID 20828914
- [Background] Bobrow BJ, Spaite DW, Berg RA, Stolz U, Sanders AB, Kern KB, Vadeboncoeur TF, Clark LL, Gallagher JV, Stapczynski JS, LoVecchio F, Mullins TJ, Humble WO, Ewy GA. Chest compression-only CPR by lay rescuers and survival from out-of-hospital cardiac arrest. JAMA. 2010 Oct 6;304(13):1447-54. doi: 10.1001/jama.2010.1392. PMID 20924010